CLINICAL TRIAL: NCT01947881
Title: Characterization of Eyes With Diabetic Macular Edema That Show Different Treatment Response to Intravitreal Anti-VEGF (CHARTRES)
Acronym: CHARTRES
Status: Completed | Type: Observational
Sponsor: Association for Innovation and Biomedical Research on Light and Image (Other)
Responsible Party: Sponsor
Other Study IDs: 4C-2013-05
Record Dates: First submitted 2013-09-17; First posted 2013-09-23 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema
Keywords: Diabetic Macular Edema; anti-VEGF; Treatment Response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with DME: Patients with DME who need treatment with anti-VEGF injections of Lucentis.

SUMMARY:
The purpose of this study is to identify Diabetic Macular Edema (DME) characteristics in eyes that show different response to treatment with anti-VEGF (vascular endothelial growth factor) injections of Lucentis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with 40 years of age or older.
* Type 2 Diabetes Mellitus.
* Glycosylated hemoglobin (HbA1C) ≤ 12% at screening visit.
* Presence of clinically significant DME involving the center (fovea) diagnosed in at least one eye that is eligible for anti-VEGF treatment in the opinion of the investigator. If both eyes are eligible, the one with the worse visual acuity, as assessed at screening visit, will be selected as the study eye.
* Visual impairment due to DME with BCVA ≥ 39 letters and ≤ 73 letters (≥ 20/160 and ≤ 20/40).
* Central subfield thickness ≥ 300µm.

Exclusion Criteria:

* Presence of any other ocular disease than DME in the study eye that may confound study results, such as Proliferative Retinopathy.
* Previous treatment with vitrectomy or intravitreous injections of triancinolone or anti-VEGF drugs in the study eye.
* Any previous laser photocoagulation (panretinal or focal) in the study eye within 6 months prior to inclusion in this study.
* Active intraocular inflammation (grade trace or above) in either eye at screening visit.
* Any active infection (e.g. conjunctivitis, keratitis, scleritis, uveitis, endophthalmitis) in either eye at screening visit.
* Important refractive errors (myopia > 6D) or opacification of clear media that interferes with images evaluation.
* Patients with renal failure or other systemic conditions which, in the opinion of the investigator, would preclude schedule study visits, completion of the study or a safe administration of study medication.
* Other criteria that in the opinion of the investigator should condition the evaluation purposed.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic Type 2 patients with clinically significant Diabetic Macular Edema with therapeutic indication for treatment with intravitreal injections of anti-VEGF Lucentis.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2014-01; Primary Completion 2015-02 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Central Retinal Thickness (Change from screening) | Change from Screening at 3 Months
  Measured by Spectral Domain Optical Coherence Tomography (OCT)
Presence of OCT diffuse macular edema (without cyst formation) (change from screening) | Change from Screening at 3 Months
Presence of neurosensorial retinal detachment. (change from screening) | Change from Screening at 3 Months
Degree of integrity of the photoreceptors in the inner/outer segments layer in the 1 mm centered in the fovea (change from screening) | Change from Screening at 3 Months
Presence and extension of capillary occlusion (change from screening) | Change from Screening at 3 Months
Area of macular leakage (intraretinal fluid volume and retinal thickness) (change frmo screening) | Change from Screening at 3 Months

SECONDARY OUTCOMES:
Best Corrected Visual Acuity (BCVA) (Change from screening) | Change from Screening at 3 Months
Central Retinal Thickness (change from screening) | Change from Screening at 6 Months
  Measured by Spectral Domain Optical Coherence Tomography (OCT)
Presence (and location) of cysts in the retinal layers (change from screening) | Change from Screening at 6 Months
Presence of OCT diffuse macular edema (without cyst formation) (change from screening) | Change from Screening at 6 months
Presence of neurosensorial retinal detachment. (change from screening) | Change from Screening at 6 Months
Degree of integrity of the photoreceptors in the inner/outer segments layer in the 1 mm centered in the fovea (change from screening) | Change from Screening at 6 months
Presence and extension of capillary occlusion (change from screening) | Change from Screening at 6 Months
Area of macular leakage (intraretinal fluid volume and retinal thickness) (change from screening) | Change from Screening at 6 Months
Best Corrected Visual Acuity (change from screening) | Change from Screening at 6 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Clinical Trials - Association for Innovation and Biomedical Research on Light and Image, Coimbra, Portugal